CLINICAL TRIAL: NCT04402437
Title: Utilization of Quadratus Lumborum Versus Lumbar Plexus Blocks for Postoperative Analgesia Following Hip Arthroplasty: A Prospective, Randomized Clinical Trial
Brief Title: QL vs LP Blocks for Analgesia Following THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Sylvia Wilson, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00098482
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Surgery

STUDY DESIGN:
Intervention Model Description: The subject will be positioned in the lateral decubitus position with the operative side up and pulse oximetry and blood pressure cuff placed for monitoring. As part of routine care, the subject will receive sedation for their comfort. All subjects would receive 20 ml of 0.5% ropivacaine in their nerve block regardless of randomization. The relevant anatomy will then be identified using either surface landmarks (lumbar plexus block) or an ultrasound (quadratus lumborum block). Surface anatomy will be marked with a marking pen for both groups to keep the intraoperative and surgical team blinded. The skin will be cleaned with chlorhexidine.
Who Masked: Participant
Masking Description: All subjects will be positioned, prepped and sedated for the randomized regional anesthesia procedure in the preoperative holding area. The subject will be positioned in the lateral decubitus position with the operative side up and pulse oximetry and blood pressure cuff placed for monitoring. As part of routine care, the subject will receive sedation for their comfort. All subjects would receive 20 ml of 0.5% ropivacaine in their nerve block regardless of randomization. The relevant anatomy will then be identified using either surface landmarks (lumbar plexus block) or an ultrasound (quadratus lumborum block). Surface anatomy will be marked with a marking pen for both groups to keep the intraoperative and surgical team blinded. The skin will be cleaned with chlorhexidine. Subject, surgeon, intraoperative anesthesia team and data collectors would all be blinded to the allocated group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receives LP Block (Active Comparator): Subjects randomized to the lumbar plexus block group will receive a subcutaneous lidocaine skin wheal 3-4 cm lateral to midline on the operative side along the intercristal line. A nerve stimulator will be sent to 1-1.5mA and a stimulating needle inserted perpendicular to the skin. The needle will be advanced slowly until the quadriceps muscle is stimulated and maintained at less than 0.6mAs. Ropivacaine (20ml, 0.5%) will be injected slowly with frequent aspiration to rule out inadvertent intravascular needle placement.
  Interventions: Procedure: LP Block
- Receives QL Block (Active Comparator): Subjects randomized to the quadratus plexus block group will receive a subcutaneous lidocaine skin wheal that will be placed after ultrasound identification of external oblique, internal oblique, transverse abdominus and quadratus lumborum muscles. A needle will then be advanced under ultrasound guidance below the internal oblique aponeurosis and lateral to the quadratus lumborum muscle. Ropivacaine (20ml, 0.5%) will be injected slowly with frequent aspiration to rule out inadvertent intravascular needle placement. Local anesthetic injection will also be observed with real time ultrasound guidance.
  Interventions: Procedure: QL Block

INTERVENTIONS:
Procedure: LP Block — Subjects randomized to the lumbar plexus block group will receive a subcutaneous lidocaine skin wheal 3-4 cm lateral to midline on the operative side along the intercristal line. A nerve stimulator will be sent to 1-1.5mA and a stimulating needle inserted perpendicular to the skin. The needle will be advanced slowly until the quadriceps muscle is stimulated and maintained at less than 0.6mAs. Ropivacaine (20ml, 0.5%) will be injected slowly with frequent aspiration to rule out inadvertent intravascular needle placement.
  Arms: Receives LP Block
Procedure: QL Block — Subjects randomized to the quadratus plexus block group will receive a subcutaneous lidocaine skin wheal that will be placed after ultrasound identification of external oblique, internal oblique, transverse abdominus and quadratus lumborum muscles. A needle will then be advanced under ultrasound guidance below the internal oblique aponeurosis and lateral to the quadratus lumborum muscle. Ropivacaine (20ml, 0.5%) will be injected slowly with frequent aspiration to rule out inadvertent intravascular needle placement. Local anesthetic injection will also be observed with real time ultrasound guidance.
  Arms: Receives QL Block

SUMMARY:
Purpose: Evaluate difference in postoperative opioid consumption when subjects receive a quadratus lumborum (QL) or lumbar plexus (LP) block preoperatively for total hip arthroplasty (THA).

Hypothesis: Preoperative QL and LP blocks will result in similar postoperative opioid consumption following hip arthroplasty.

DETAILED DESCRIPTION:
With the goal of improving physical function and quality of life, the demand for total hip arthroplasty (THA) continues to grow. However, postoperative pain associated with THA remains a serious concern for patients. In the middle of a growing opioid epidemic, multimodal approaches utilizing both non-opioid analgesics and regional anesthetic techniques are being increasingly sought.

Regional anesthetic techniques are associated with both decreased opioid consumption and pain scores compared with systemic analgesia alone. However, regional techniques for THA are seldom compared. Lumbar plexus blocks are commonly performed for postoperative analgesia for THA. However, more recent case reports have described utilizing quadratus lumborum blocks for analgesia following hip fracture and THA.

This prospective study would randomize subjects to receive a lumbar plexus block or quadratus lumborum block prior to THA. The primary end point would be opioid consumption at 12 hours postoperative. Our hypothesis is that opioid consumption will not differ between groups.

The quadratus lumborum block is a fascial plane block. Originally described for abdominal surgery, numerous case reports and editorial publications have highlighted the effectiveness of quadratus lumborum (QL) blocks as an analgesic technique for hip fracture and hip arthroplasty. However, prospective randomized studies comparing QL blocks to other regional techniques for THA analgesia are lacking.

The lateral approach to the QL block is performed by injecting local anesthetic deep to the transversus abdominus abdominus apnoneurosis and superficial to the fascia transversalis with direct ultrasound guidance. After completing consent, placing monitors and providing mild sedation, the subject is positioned laterally and the muscular anatomy (external oblique, internal oblique, transverse abdominis, quadratus lumborum and latissimus dorsi muscles) identified. After placing a subcutaneous skin wheal with lidiocaine, a blunt regional anesthesia needle is inserted using in-plane ultrasound guidance. Local anesthetic is deposited incrementally with frequent aspiration in the anterolateral border of the quadratus lumborum muscle at the junction of the transversalis fascia, outside the anterior layer of the thoracolumbar fascia and superficial to the fascia transversalis.

Risks of anterior approach to the quadratus lumborum block are similar to most truncal blocks and include infection, bleeding, bowel perforation or local anesthetic toxicity (LAST). Infection risk is minimized by utilizing appropriate antiseptic and sterile technique as is standard for any regional procedure. Risk of a retroperitoneal hematoma is increased with the posterior approach to the quadratus lumborum block because of its transmuscular approach and likelihood of abdominal branches of lumbar arteries in the path of the needle. For this reason, the posterior approach to the quadratus lumborum block will not be used for this study. The risk of LAST is a risk with any regional procedure and is minimized by frequent aspiration, incremental local anesthetic injection and vital signs monitoring throughout.

The quadratus lumborum block is already a block utilized for a variety of surgical procedures to decrease postoperative pain. Potential benefits to the QL block over the common lumbar plexus block include more superficial block placement and ultrasound visualization. The investigator hypothesize that preoperative QL blocks will reduce opioid consumption similar to lumbar plexus blocks following elective hip arthroplasty.

Information regarding the study will be presented to subjects in the surgical clinic or preoperative anesthesia clinic in the preoperative period. Subjects will be educated on the role of regional anesthesia in postoperative analgesia. Subjects will be able to consider the study until the day of surgery. On the day of surgery, subjects may then choose to provide written consent or decline to participate.

Subjects will be enrolled on the day of surgery in the preoperative holding area.

After discussion in the preoperative holding area regarding risks and benefits of both the lumbar plexus and QL block, subjects will be consented if they choose to participate. Consent will be obtained from subject by an IRB approved CITI certified study team member that has been trained on the protocol. Written consent with a witness will be completed once all questions are answered and exclusion and inclusion verified. Copies of all documents will be provided to the subjects. Once subjects are consented, they will be assigned an enrollment number. Prior to subject enrollment, randomization will done by a statistician and randomized group (lumbar plexus block (current practice) or QL block) assigned based on the subject enrollment number.

Design: This prospective, single blinded clinical trial will randomize subject to receive a lumbar plexus or QL block prior to THA. The randomization will be created by a statistician prior to subject enrollment.

Groups: Subjects will be randomized to receive a preoperative lumbar plexus (n = 100) or QL (n = 100 ) block prior to THA.

Potential participants that are on the operating room schedule for THA will be screened for eligibility via chart review.

Once subjects have signed an informed consent, they will be assigned an enrollment number. Numbers would be assigned sequentially with the first enrolled subject receiving "001," the second subject receiving "002," and the last subject receiving number "184." Randomization will be created prior to the study starting by a statistician with half of the research subject number being assigned to receive a QL block and the other half assigned to receive a lumbar plexus block, which is our current standard of care. The regional anesthesia team will open the envelope labeled with the subject's assigned number to reveal the randomization.

Following informed consent, all subjects will be positioned, prepped and sedated for the randomized regional anesthesia procedure in the preoperative holding area. The subject will be positioned in the lateral decubitus position with the operative side up and pulse oximetry and blood pressure cuff placed for monitoring. As part of routine care, the subject will receive sedation for their comfort. All subjects would receive 20 ml of 0.5% ropivacaine in their nerve block regardless of randomization. The relevant anatomy will then be identified using either surface landmarks (lumbar plexus block) or an ultrasound (quadratus lumborum block). All participants, regardless of group assignment, will be positioned, have an area on their back and side cleaned, have an ultrasound placed, and numbing medication placed just below the skin at both block sites (skin wheal). This will be done so that participant and the team collecting result will be blinded. Subject, surgeon, intraoperative anesthesia team and data collectors would all be blinded to the allocated group.

Subjects randomized to the lumbar plexus block group will receive a subcutaneous lidocaine skin wheal 3-4 cm lateral to midline on the operative side along the intercristal line. A nerve stimulator will be sent to 1-1.5mA and a stimulating needle inserted perpendicular to the skin. The needle will be advanced slowly until the quadriceps muscle is stimulated and maintained at less than 0.6mAs. Ropivacaine (20ml, 0.5%) will be injected slowly with frequent aspiration to rule out inadvertent intravascular needle placement.

Subjects randomized to the quadratus plexus block group will receive a subcutaneous lidocaine skin wheal that will be placed after ultrasound identification of external oblique, internal oblique, transverse abdominus and quadratus lumborum muscles. A needle will then be advanced under ultrasound guidance below the internal oblique aponeurosis and lateral to the quadratus lumborum muscle. Ropivacaine (20ml, 0.5%) will be injected slowly with frequent aspiration to rule out inadvertent intravascular needle placement. Local anesthetic injection will also be observed with real time ultrasound guidance.

The participant's chart will be reviewed for data collection.

Participants will also be asked to perform a Visual Analog Scale pain score preoperatively (baseline), postoperatively (once awake) and approximately 24 hours post operatively.

Care in the perioperative period will otherwise be standardized. In the post-anesthesia care unit (PACU), hydromorphone or morphine will be titrated by the PACU nurse for the subject's comfort.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years-old
* Undergoing elective hip arthroplasty.

Exclusion Criteria:

* Local anesthetic allergy
* Chlorhexidine allergy
* Subjects with a weight less than 40kg
* Subjects that are unable or choose not to give informed consent
* Emergency surgery
* Known preoperative substance abuse
* Allergy to all opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 12 hours
  Opioid consumption including intraoperative consumption

SECONDARY OUTCOMES:
Opioid consumption 8 hours postoperative | 8 hours
  Opioid consumption including intraoperative consumption

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia H Wilson, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Bruyere O, Ethgen O, Neuprez A, Zegels B, Gillet P, Huskin JP, Reginster JY. Health-related quality of life after total knee or hip replacement for osteoarthritis: a 7-year prospective study. Arch Orthop Trauma Surg. 2012 Nov;132(11):1583-7. doi: 10.1007/s00402-012-1583-7. Epub 2012 Jul 28. PMID 22842917
- [Background] Ethgen O, Bruyere O, Richy F, Dardennes C, Reginster JY. Health-related quality of life in total hip and total knee arthroplasty. A qualitative and systematic review of the literature. J Bone Joint Surg Am. 2004 May;86(5):963-74. doi: 10.2106/00004623-200405000-00012. PMID 15118039
- [Background] Singh JA, Lewallen D. Predictors of pain and use of pain medications following primary Total Hip Arthroplasty (THA): 5,707 THAs at 2-years and 3,289 THAs at 5-years. BMC Musculoskelet Disord. 2010 May 13;11:90. doi: 10.1186/1471-2474-11-90. PMID 20462458
- [Background] Becchi C, Al Malyan M, Coppini R, Campolo M, Magherini M, Boncinelli S. Opioid-free analgesia by continuous psoas compartment block after total hip arthroplasty. A randomized study. Eur J Anaesthesiol. 2008 May;25(5):418-23. doi: 10.1017/S026502150700302X. Epub 2007 Nov 21. PMID 18028577
- [Background] Biboulet P, Morau D, Aubas P, Bringuier-Branchereau S, Capdevila X. Postoperative analgesia after total-hip arthroplasty: Comparison of intravenous patient-controlled analgesia with morphine and single injection of femoral nerve or psoas compartment block. a prospective, randomized, double-blind study. Reg Anesth Pain Med. 2004 Mar-Apr;29(2):102-9. doi: 10.1016/j.rapm.2003.11.006. PMID 15029544
- [Background] Macfarlane AJ, Prasad GA, Chan VW, Brull R. Does regional anaesthesia improve outcome after total hip arthroplasty? A systematic review. Br J Anaesth. 2009 Sep;103(3):335-45. doi: 10.1093/bja/aep208. Epub 2009 Jul 23. PMID 19628483
- [Background] Stevens RD, Van Gessel E, Flory N, Fournier R, Gamulin Z. Lumbar plexus block reduces pain and blood loss associated with total hip arthroplasty. Anesthesiology. 2000 Jul;93(1):115-21. doi: 10.1097/00000542-200007000-00021. PMID 10861154
- [Background] Harvey NR, Wolf BJ, Bolin ED, Wilson SH. Comparison of analgaesia with lumbar epidurals and lumbar plexus nerve blocks in patients receiving multimodal analgaesics following primary total hip arthroplasty: a retrospective analysis. Int Orthop. 2017 Nov;41(11):2229-2235. doi: 10.1007/s00264-017-3465-7. Epub 2017 Apr 11. PMID 28396932
- [Background] Wilson SH, Wolf BJ, Algendy AA, Sealy C, Demos HA, McSwain JR. Comparison of Lumbar Epidurals and Lumbar Plexus Nerve Blocks for Analgesia Following Primary Total Hip Arthroplasty: A Retrospective Analysis. J Arthroplasty. 2017 Feb;32(2):635-640. doi: 10.1016/j.arth.2016.07.042. Epub 2016 Aug 10. PMID 27597428
- [Background] Wilson SH, Auroux AS, Eloy JD, Merman RB, Chelly JE. Ropivacaine 0.1% versus 0.2% for continuous lumbar plexus nerve block infusions following total hip arthroplasty: a randomized, double blinded study. Pain Med. 2014 Mar;15(3):465-72. doi: 10.1111/pme.12309. Epub 2013 Dec 11. PMID 24330381
- [Background] Hockett MM, Hembrador S, Lee A. Continuous Quadratus Lumborum Block for Postoperative Pain in Total Hip Arthroplasty: A Case Report. A A Case Rep. 2016 Sep 15;7(6):129-31. doi: 10.1213/XAA.0000000000000363. PMID 27513972
- [Background] Johnston DF, Sondekoppam RV. Continuous quadratus lumborum block analgesia for total hip arthroplasty revision. J Clin Anesth. 2016 Dec;35:235-237. doi: 10.1016/j.jclinane.2016.08.002. Epub 2016 Sep 26. No abstract available. PMID 27871532
- [Background] La Colla L, Ben-David B, Merman R. Quadratus Lumborum Block as an Alternative to Lumbar Plexus Block for Hip Surgery: A Report of 2 Cases. A A Case Rep. 2017 Jan 1;8(1):4-6. doi: 10.1213/XAA.0000000000000406. PMID 28036319
- [Background] La Colla L, Uskova A, Ben-David B. Single-shot Quadratus Lumborum Block for Postoperative Analgesia After Minimally Invasive Hip Arthroplasty: A New Alternative to Continuous Lumbar Plexus Block? Reg Anesth Pain Med. 2017 Jan/Feb;42(1):125-126. doi: 10.1097/AAP.0000000000000523. No abstract available. PMID 27997495
- [Background] Ueshima H, Yoshiyama S, Otake H. RETRACTED: The ultrasound-guided continuous transmuscular quadratus lumborum block is an effective analgesia for total hip arthroplasty. J Clin Anesth. 2016 Jun;31:35. doi: 10.1016/j.jclinane.2015.12.033. Epub 2016 Mar 22. PMID 27185672 (Retraction: PMID 35393191 J Clin Anesth. 2022 Aug;79:110702; PMID 35397960 J Clin Anesth. 2022 Aug;79:110704)
- [Background] Hansen CK, Dam M, Bendtsen TF, Borglum J. Ultrasound-Guided Quadratus Lumborum Blocks: Definition of the Clinical Relevant Endpoint of Injection and the Safest Approach. A A Case Rep. 2016 Jan 15;6(2):39. doi: 10.1213/XAA.0000000000000270. No abstract available. PMID 26771297
- [Background] Capdevila X, Macaire P, Dadure C, Choquet O, Biboulet P, Ryckwaert Y, D'Athis F. Continuous psoas compartment block for postoperative analgesia after total hip arthroplasty: new landmarks, technical guidelines, and clinical evaluation. Anesth Analg. 2002 Jun;94(6):1606-13, table of contents. doi: 10.1097/00000539-200206000-00045. PMID 12032037
- [Derived] Kelly T, Wolla CD, Wolf BJ, Hay E, Babb S, Wilson SH. Comparison of lateral quadratus lumborum and lumbar plexus blocks for postoperative analgesia following total hip arthroplasty: a randomized clinical trial. Reg Anesth Pain Med. 2022 Sep;47(9):541-546. doi: 10.1136/rapm-2022-103598. Epub 2022 Jun 10. PMID 35688515